CLINICAL TRIAL: NCT02145364
Title: Evaluation of the Ulthera® System for Correction of Moderate to Severe Atrophic Acne Scars
Brief Title: Ultherapy® for the Treatment of Acne Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ULT-139
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Last update posted 2017-12-14 (Actual); Status verified 2015-10

CONDITIONS: Acne Scars; Atrophic Acne Scars
Keywords: Ulthera System®; Ultherapy®; Ulthera, Inc.

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ultherapy® treatment of acne scars (Experimental): Subjects receiving dual depth treatment of acne scars using the 7MHz,3.0mm and 10MHz,1.5mm transducers.
  Interventions: Device: Ultherapy® treatment

INTERVENTIONS:
Device: Ultherapy® treatment — Microfocused ultrasound treatment
  Other Names: Ulthera System®

SUMMARY:
This is a prospective, multi-site trial to be conducted at 2 clinical sites. Up to 20 subjects will receive study treatments. Following study treatments, follow-up visits will occur at 60, 90 and 180 days from each subject's last study treatment.

DETAILED DESCRIPTION:
Subjects with moderate to severe atrophic acne scars will be enrolled. Subjects will receive up to three dual-depth treatments to the cheek and temple areas impacted by acne scars, treating the number of treatment squares necessary to cover the area of scarring. Each treatment square will receive 30 lines per transducer depth for a total of 60 lines per treatment square. Three treatments 30 days apart will be required.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 to 70 years.
* Subject in good health.
* Presence of moderate to severe atrophic acne scars on the cheeks and/or temples.
* Scars must be rolling and boxcar type scars predominantly, with few to no icepick scars present.
* Scars should be distensible with tension applied to skin.
* Subject must desire correction of his/her acne scarring as demonstrated by any level of dissatisfaction on baseline PSQ.
* Subjects of all Fitzpatrick skin types are eligible.
* Subject must be willing to withhold additional aesthetic therapies in the areas to be treated for the entire study duration if these treatments are judged by the investigator to potentially impact results.
* Willingness and ability to comply with protocol requirements, including returning for follow-up visits
* Willingness to maintain current skin care regimen and refrain from adding any new products or drugs for acne or acne scars for the duration of the study.
* Subjects of childbearing potential must have a negative urine pregnancy test result and must not be lactating at the Screening Visit and be willing and able to use an acceptable method of birth control during the study.
* Absence of physical or psychological conditions unacceptable to the investigator.
* Willingness and ability to provide written consent for study-required photography and adherence to photography procedures.
* Willingness and ability to provide written informed consent and HIPAA authorization prior to performance of any study-related procedure.

Exclusion Criteria:

* Presence of an active systemic or local skin disease that may affect wound healing.
* Severe solar elastosis.
* Recent history of significant trauma to the face (<6 months).
* Significant scarring, other than acne scars in area(s) to be treated.
* Open wounds or lesions in the area(s) to be treated.
* Severe or cystic active and clinically significant acne on the area(s) to be treated.
* Have a recent or current history of inflammatory skin disease, infection, cancerous/pre-cancerous lesion, unhealed wound in the proposed treatment areas.
* Have a history of systemic granulomatous diseases active or inactive or connective tissue disease.
* Have hypertrophic acne scars, any evidence of keloid scarring, predominantly icepick scarring (defined as more than half of all scar area in either the left or right or treatment area) or sinus tract scars.
* Presence of a metal stent or implant in the area(s) to be treated.
* Inability to understand protocol or give informed consent.
* Microdermabrasion or glycolic acid peels to the treatment area(s) within four weeks prior to study participation or during the study.
* History of allergic reaction to Ibuprofen, Acetaminophen, or Lidocaine/Tetracaine.
* History of chronic drug or alcohol abuse.
* History of autoimmune disease.
* Concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study device.
* Subjects who anticipate the need for surgery or overnight hospitalization during the study.
* Subjects who, in the investigator's opinion, have a history of poor cooperation, noncompliance with medical treatment, or unreliability.
* Concurrent enrollment, or participated within the past 30 days, in any study involving the use of investigational devices or drugs.
* Current smoker or history of smoking in the last two years.
* History of the following cosmetic treatments in the areas to be treated:

  1. Skin tightening procedure within the past year;
  2. Injectable filler of any type within the past: i. 12 months for Hyaluronic acid fillers (e.g.,Restylane); ii. 12 months for Ca Hydroxyapatite fillers (e.g., Radiesse); iii. 24 months for Poly-L-Lactic acid fillers (e.g., Sculptra); iv. Cultured fibroblast (e.g. LaViv) within the past two years; v. Ever for permanent fillers (e.g., Silicone, ArteFill)
  3. Neurotoxins within the past three months;
  4. Ablative resurfacing laser treatment within the past two years;
  5. Nonablative, rejuvenative laser or light treatment within the past six months;
  6. Surgical dermabrasion or deep facial peels within the past two years;
  7. Any history of contour threads.
* History of using the following prescription medications

  1. Accutane or other systemic retinoids within the past six months;
  2. Topical retinoids within the past two weeks;
  3. Antiplatelet agents / Anticoagulants (Coumadin, Heparin, Plavix, chronic NSAID use);
  4. Aspirin greater than 82mg/day
  5. Psychiatric drugs that in the investigators opinion would impair the subject from understanding the protocol requirements or understanding and signing the informed consent or affect their ability to accurately complete QOL and subjective improvement assessments.
* Any condition which in the opinion of the investigator makes the patient unable to complete the study per protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-05; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Acne Scar Improvement Scale | 90 Days post-treatment #3
  Determined by a masked, qualitative assessment of photographs at 90 days post final treatment compared to baseline. Clinical improvement will be assessed by the investigator from the visual of the treated area according to the following scale: -1 for exacerbation, 0 no change, 1 for 1%-25% improvement, 2 for 25%-50% improvement, 3 for 50%-75% improvement, and 4 for 75%-99% improvement.
Acne Scar Improvement Scale | 180 days post-treatment #3
  Determined by a masked, qualitative assessment of photographs at 180 days post final treatment compared to baseline. Clinical improvement will be assessed by the investigator from the visual of the treated area according to the following scale: -1 for exacerbation, 0 no change, 1 for 1%-25% improvement, 2 for 25%-50% improvement, 3 for 50%-75% improvement, and 4 for 75%-99% improvement.

SECONDARY OUTCOMES:
Physician Scar Improvement Scale (PSIS) and Self-Assessed Scar Improvement Scale (SASIS) | 60 days post-treatment #3
  Determined by PSIS (clinician) assessment and SASIS (subject) assessment at 60 days post final treatment compared to baseline. Clinical improvement will be assessed from the visual assessment of the treated area according to the following scale: -1 for exacerbation, 0 no change, 1 for 1%-25% improvement, 2 for 25%-50% improvement, 3 for 50%-75% improvement, and 4 for 75%-99% improvement.
Physician Scar Improvement Scale (PSIS) and Self-Assessed Scar Improvement Scale (SASIS) | 90 days post-treatment #3
  Determined by PSIS (clinician) assessment and SASIS (subject) assessment at 90 days post final treatment compared to baseline. Clinical improvement will be assessed from the visual assessment of the treated area according to the following scale: -1 for exacerbation, 0 no change, 1 for 1%-25% improvement, 2 for 25%-50% improvement, 3 for 50%-75% improvement, and 4 for 75%-99% improvement.
Physician Scar Improvement Scale (PSIS) and Self-Assessed Scar Improvement Scale (SASIS) | 180 days post-treatment #3
  Determined by PSIS (clinician) assessment and SASIS (subject) assessment at 180 days post final treatment compared to baseline. Clinical improvement will be assessed from the visual assessment of the treated area according to the following scale: -1 for exacerbation, 0 no change, 1 for 1%-25% improvement, 2 for 25%-50% improvement, 3 for 50%-75% improvement, and 4 for 75%-99% improvement.
Physician Acne Scar Assessment Scale | 60 days post-treatment #3
  Severity of acne scarring is are graded on a 5-point scale (0-4), where 0 = clear, 1= very mild, 2= mild, 3= moderate, 4= severe, comparing the grade assessed at 60 days following the final study treatment to the baseline grade.
Physician Acne Scar Assessment Scale | 90 days post-treatment #3
  Severity of acne scarring is are graded on a 5-point scale (0-4), where 0 = clear, 1= very mild, 2= mild, 3= moderate, 4= severe, comparing the grade assessed at 90 days following the final study treatment to the baseline grade.
Physician Acne Scar Assessment Scale | 180 days post-treatment #3
  Severity of acne scarring is are graded on a 5-point scale (0-4), where 0 = clear, 1= very mild, 2= mild, 3= moderate, 4= severe, comparing the grade assessed at 180 days following the final study treatment to the baseline grade.
Clinician Global Aesthetic Improvement Scale (CGAIS) and Subject Global Aesthetic Improvement Scale (SGAIS) | 60 days post-treatment #3
  Overall aesthetic improvement assessed based on a live assessment of the subject and a photographic assessment comparing 60 day post-treatment photos to baseline photos. The GAIS is a 5-point scale (1-5) describing an overall assessment as follows:
  1. - Very Much Improved
  2. - Much Improved
  3. - Improved
  4. - No Change
  5. - Worse
Clinician Global Aesthetic Improvement Scale (CGAIS) and Subject Global Aesthetic Improvement Scale (SGAIS) | 90 days post-treatment #3
  Overall aesthetic improvement assessed based on a live assessment of the subject and a photographic assessment comparing 90 day post-treatment photos to baseline photos. The GAIS is a 5-point scale (1-5) describing an overall assessment as follows:
  1. - Very Much Improved
  2. - Much Improved
  3. - Improved
  4. - No Change
  5. - Worse
Clinician Global Aesthetic Improvement Scale (CGAIS) and Subject Global Aesthetic Improvement Scale (SGAIS) | 180 days post-treatment #3
  Overall aesthetic improvement assessed based on a live assessment of the subject and a photographic assessment comparing 180 day post-treatment photos to baseline photos. The GAIS is a 5-point scale (1-5) describing an overall assessment as follows:
  1. - Very Much Improved
  2. - Much Improved
  3. - Improved
  4. - No Change
  5. - Worse
Patient Satisfaction Questionnaire (PSQ) | 90 days post-treatment #3
  Patient satisfaction determined by scores on a PSQ completed at 90 days post-treatment #3, indicating improvement in the areas treated and characterizing satisfaction with study treatment, i.e., Extremely Satisfied, Satisfied, Slightly Satisfied, Neither Satisfied or Dissatisfied, Slightly Dissatisfied, Dissatisfied, Extremely Dissatisfied.

CONTACTS AND LOCATIONS:
Overall Officials: John Joseph, MD, Principal Investigator — Clinical Testing of Beverly Hills; Corey Maas, MD, Principal Investigator — The Maas Clinic
Locations (2):
- United States (2):
  - Clinical Testing of Beverly Hills, Beverly Hills, California
  - The Maas Clinic, San Francisco, California